CLINICAL TRIAL: NCT05115162
Title: The Effects of the Hybrid Telerehabilitation Exercise Program in Inactive University Students During Covid-19 Pandemic - A Randomized Controlled Study
Brief Title: The Effects of the Hybrid Telerehabilitation Exercise in Inactive Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2021.170
Record Dates: First submitted 2021-11-01; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Physical Activity; Exercise
Keywords: Hybrid Telerehabilitation; Sleep Quality; Depression; Physical Inactivity; Exercise
MeSH Terms: conditions — Motor Activity; Sleep Initiation and Maintenance Disorders; Depression; Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- elerehablitation home exercise group (Experimental): Telerehabilitation home exercise group received indoor walking and general exercise program for 6 weeks.
  Indoor walking was performed 3 days a week, for 30 minutes. General exercise program was consisted of flexibility, strengthening the shoulder and trunk muscles, bridge exercises, lying on the back, cycling and squatting exercises. All of the general exercises were repeated 3 days a week, 2 sets and each set with 10 repetitions.
  Two synchronized exercise education sessions were performed with the exercise group. In the first of these sessions, the content of the exercise program was explained. In the second, it was checked whether the exercises were done correctly. After synchronous education sessions, an asynchronous home exercise program, consisting walking and general exercise program continued for 6 weeks.
  Interventions: Other: Exercise
- Control Group (No Intervention): This group did not participate in any exercise program for 6 weeks.

INTERVENTIONS:
Other: Exercise — The exercises consist of flexibility, strengthening exercises for the trunk and extremities, and walking indoors.The walking program was applied for at least 30 minutes. Eight different exercises were given for the trunk and extremities and these exercises were applied 3 times a week, 2 sets, each set with 10 repetitions.
  Arms: elerehablitation home exercise group

SUMMARY:
The aim of this study was to examine the effects of a 6-week hybrid telerehabilitation exercise program on sleep quality, depression and quality of life of university students with physical inactivity.

DETAILED DESCRIPTION:
COVID-19 pandemic have caused multidimensional effects on people of all ages. Technology-based applications are widely using especially in education and health systems. The use of telerehabilitation services scope expanded throughout the pandemic. Precautions such as curfews and closing sports halls due to the pandemic have increased the time that being physically inactive in individuals. Since higher education continues with online systems and continuing stay home politics, positive or negative changes occurred in the lifestyles of students. It was shown activity, sleep, and psychological problems in young population. This problems are important because of their serious effects and comorbities, on pain, posture, and muscles. Exercise, sleep quality and quality of life are associated with each other a major proportion. Since inactivity and pandemic precautions, university students' quality of life and social life was disturbed negatively. On the other hand attendance the physical activity and exercise are important protective method for these negative situations. Therefore, this study planned to investigate the effects of home exercise program performed with the telerehabilitation method on sleep, depression, and quality of life on undergraduate students in the Covid-19 outbreak.

The population sample of the study consists of healthy sedentary individuals in the 18-65 age group. Gpower 3.1.9.7 software was used while calculating the sample size to be included in the study. The alpha error was 5%, the power of the study was 80%, and the effect size was 0.8. As a result of this calculation, taking into account the possibility of participants leaving the program, a total of 86 participants were included in the study and the study was completed with 63 people. Participants were randomly divided into 2 groups as 32 exercise group and 31 control group. Internet-based software (www.randomizer.org) was used for randomization. Both groups were evaluated at the beginning of the study and after 6 weeks. The exercise program was applied for 6 weeks. The exercises were repeated 3 days a week, 2 sets and each set with 10 repetitions. Two synchronized sessions were performed with the exercise group. In the first of these sessions, the content of the exercise program was explained. In the second, it was checked whether the exercises were done correctly. There were 3 days between synchronized sessions. No program was applied to the control group for 6 weeks, but at the end of the study, the same exercises given to the exercise group were also shown to the control group.

Exercise program consisted of indoor walking (30-minutes), flexibility, strengthening the shoulder and trunk muscles, bridge exercises, lying on the back, cycling and squatting.

Statistical Analysis: Independent Sample T Test was used to compare data with normal distribution between groups. To inter-group analysis, Paired Sample T Test was used and significance level was accepted as <0.05.

ELIGIBILITY:
Inclusion Criteria:

* ....>18 years old
* Pittsburg Sleep Quality Index total score >5 points
* No history of orthopedic, neurological, or cardiovascular disease
* Physical activity level < 600 MET-min-week according to International Physical Activity Questionnaire-Short From.
* Cooperative
* Not exposed to any telerehabilitation application

Exclusion Criteria:

* Having cancer, diabetes mellitus, pregnancy, infection, rheumatic pain
* Less than 85% attendance to the program
* Participating in any other physical activity program

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-01-17 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI): | At the baseline
  Measurement of the sleep quality
Pittsburgh Sleep Quality Index | At the end of the 6th week
  Measurement of the sleep quality

SECONDARY OUTCOMES:
Beck Depression Inventory | At the baseline
  Measurement of the depression level
Beck Depression Inventory | At the end of the 6th week
  Measurement of the depression level
Short Form-12 | At the baseline
  Measurement of the quality of life
Short Form-12 | At the end of the 6th week
  Measurement of the quality of life
International Physical Activity Questionnaire-Short Form | At the baseline
  Measurement of the physical activity
International Physical Activity Questionnaire-Short Form | At the end of the 6th week
  Measurement of the physical activity
Adherence the exercise program | At the end of the 6th week
  Attendance to the exercise program (for exercise group). It was calculated at the end of the 6th week according to the percentage of completing the exercise sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No